CLINICAL TRIAL: NCT06386770
Title: Systemic Versus Local Dexamedetomedine as An Adjuvant to Bupivacaine in Ultrasound Guided Erector Spinae Block in Kidney Exploration Surgeries ,A Randomized Controlled Trial
Brief Title: Systemic Versus Local Dexmedetomidine as An Adjuvant to Bupivacaine in Ultrasound Guided Erector Spinae Block
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Soudy Salah Hammad, Lecturer of anesthesia and surgical intensive care, Aswan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Asw.U./742 /2/23
Record Dates: First submitted 2024-04-04; First posted 2024-04-26 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-05

CONDITIONS: Erector Spinae Block; Dexmedetomidine
Keywords: Bupivacaine; kidney exploration surgery
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: These prospective, randomized, controlled clinical trials will be performed in Aswan University Hospital on 75 patients who are scheduled for kidney exploration surgeries
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In our randomized controlled trial, we employed masking (also called blinding) to reduce bias. Participants were unaware of whether they were receiving the intervention or control. Caregivers were instructed not to reveal this information, and outcome assessors who evaluated results were kept separate from intervention delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group Ι Block only (group BO) (control group) (Active Comparator): Ultrasound guided erector spinae block will receive 30 ml (28 ml bupivacaine 0.25% +2ml normal saline Na cl 0,9 %) +10ml IV normal saline will be injected over 10 min after 10 min from the induction of general anesthesia
  Interventions: Drug: Bupivacaine Hydrochloride
- Group ΙI (group DL): (Active Comparator): Ultrasound guided erector spinae block will receive 30 ml (28 ml bupivacaine 0.25% plus dexmedetomidine (0.5µg/kg) diluted in 2ml normal saline Na cl 0,9%) + 10ml IV normal saline will be injected over 10 min after 10 min from the induction of general anesthesia
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Group III (group D IV): (Active Comparator): Ultrasound guided erector spinae block will receive 30 ml (28 ml bupivacaine 0.25% +2ml normal saline Na cl 0,9%) + dexmedetomidine (0.5µg/kg) diluted with 10 ml normal saline IV infusion by syringe pump over 10 min after 10 min from the induction of general anesthesia
  Interventions: Drug: Dexmedetomidine in 0.9 % NaCl 200 Mcg/50 mL (4 Mcg/mL) INTRAVEN INFUSION BOTTLE (ML)

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — Group ΙI (group DL): erector spinae block will receive 30 ml (28 ml bupivacaine 0.25% plus dexamedetomedine (0.5µg/kg) diluted in 2ml normal saline Na cl 0,9% ) + 10ml IV normal saline will be injected over 10 min after 10 min from the induction of general anesthesia
  Arms: Group ΙI (group DL):
Drug: Bupivacaine Hydrochloride — .Group Ι Block only (group BO) (control group): erector spinae block will receive 30 ml ( 28 ml bupivacaine 0.25% +2ml normal saline Na cl 0,9 %) +10ml IV normal saline will be injected over 10 min after 10 min from the induction of general anesthesia
  Arms: Group Ι Block only (group BO) (control group)
Drug: Dexmedetomidine in 0.9 % NaCl 200 Mcg/50 mL (4 Mcg/mL) INTRAVEN INFUSION BOTTLE (ML) — Group III (group D IV): erector spinea block will receive 30 ml ( 28 ml bupivacaine 0.25% +2ml normal saline Na cl 0,9%) + dexamedetomedine (0.5µg/kg) diluted with 10 ml normal saline IV infusion by syringe pump over 10 min after 10 min from the induction of general anesthesia.
  Arms: Group III (group D IV):

SUMMARY:
The aim of this study is to investigate the analgesic effect of local versus systemic dexamedetomedine as adjuvant to bupivacaine in erector spinae block in kidney exploration surgeries.

DETAILED DESCRIPTION:
Open Kidney surgeries remain one of the approaches used for those patients are requiring partial or radical nephrectomy and is associated with a high incidence of intense immediate postoperative pain and chronic pain for months following surgery.

Effective treatment of postoperative pain allows early mobilization of the patient, shortens the recovery and discharge time, prevents the development of chronic pain, and increases satisfaction and long-term quality of life.

Current modalities used to manage pain for patients undergoing kidney exploration include oral and parenteral opioid administration, local anesthetic infiltration, and certain neuraxial and regional anesthesia procedures including thoracic epidurals and paravertebral blocks.

The erector spinae plane (ESP) block is a newer regional anesthetic technique that can be used to provide analgesia for a variety of surgical procedures or to manage acute or chronic pain. The technique is relatively easy to perform on patients, and it is performable with minimal or no sedation in the pre-operative holding area.

Ultrasound is a non-invasive visualization technology that helps capture the anatomical structure of target tissues; it can help guide the direction and depth of anesthesia puncture needles, thus reducing the risk of complications.

The local anesthetic drugs have a limited duration of action, so we need to add adjuvants such as opioids, alpha two agonists, neostigmine, or magnesium.

Dexmedetomidine is a potent α2 agonist and is a powerful adjuvant to regional anesthesia and analgesia. It can prolong the duration of the nerve block anesthesia resulting in increased effectiveness of the block in terms of duration, less use of opioids, and shorter hospital stay in the absence of clinically significant side effects (hypotension, nausea, vomiting, and pruritus.

Adding adjuvants to local anesthetics is frequently used to prolong the duration of single-injection regional nerve block.

There have been multiple studies claiming increased effectiveness of use of dexmedetomidine and this has been consolidated in a meta-analysis examining the effectiveness of dexamedetomedine as a peripheral nerve block adjuvant.

ELIGIBILITY:
Inclusion Criteria:

•. kidney exploration surgeries.

* ASA I/II patients.
* BMI <35

Exclusion Criteria:

* Getting opioid analgesics prior to surgery.
* Local infections at the site where needle for block is to be inserted.
* ASAIII/IV.
* Pregnancy.
* History of drug addiction or alcohol abuse or a psychiatric illness,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The duration of analgesia, this was defined as the time in minutes to the first request for postoperative analgesics. | at 60 , 180 minutes
  The duration of analgesia, this was defined as the time in minutes to the first request for

SECONDARY OUTCOMES:
2. Total postoperative opioid consumption (Nalbuphine consumption (mg) within the 48-hour period . | at 1, 3, 6, 12, 24, 36 and 48 hours
  2. Total postoperative opioid consumption (Nalbuphine consumption (mg) within the 48-hour period.
Ramsay Sedation Scale (RSS) (1: anxious; 2: cooperative and tranquil; 3: responding to command; 4: brisk response to stimuli; 5: sluggish response to stimuli; and 6: no response to stimuli) will be all assessed | at 1, 3, 6, 12, 24, 36 and 48 hours
  amsay Sedation Scale (RSS) The RSS is a user-friendly and therefore commonly used sedation scale, with scores ranging from +4 (a violent dangerous patient) to -5 (an unarousable patient).6 A sedation score of 0 is most often therapeutically targeted, as it correlates with an alert and calm patient.
Intraoperative hemodynamic parameters blood pressure | at 1, 3, 6, hours
  blood pressure measurement obtained by non-invasive blood pressure cuff during intraoperative and postoperative in PACU expressed in mmhg
Minimum alveolar concentration (MAC) requirements | during intraoperative periods expressed in minutes
  Minimum alveolar concentration or MAC is the concentration, often expressed as a percentage by volume, of a vapour in the alveoli of the lungs that is needed to prevent movement (motor response) in 50% of subjects in response to surgical (pain) stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab A Mahmoud, MSc, Study Chair — Aswan University; Ayman M Eldemrdash, Principal Investigator — Aswan University
Locations (1):
- Aswan University, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Wang Q, Li H, Wei S, Zhang G, Ni C, Sun L, Zheng H. Dexmedetomidine Added to Ropivacaine for Ultrasound-guided Erector Spinae Plane Block Prolongs Analgesia Duration and Reduces Perioperative Opioid Consumption After Thoracotomy: A Randomized, Controlled Clinical Study. Clin J Pain. 2021 Oct 12;38(1):8-14. doi: 10.1097/AJP.0000000000000992. PMID 34636753